CLINICAL TRIAL: NCT03062111
Title: Laser Enucleation of Prostate (LEP) Versus Transurethral Resection of Prostate (TURP): a Prospective Study Comparing Outcomes
Brief Title: Laser Enucleation of Prostate (LEP) Versus Transurethral Resection of Prostate (TURP)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to low enrollment.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-36011
Record Dates: First submitted 2017-01-30; First posted 2017-02-23 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Laser Enucleation of Prostate (LEP); Transurethral Resection of Prostate (TURP)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProTouch Laser Enucleation of Prostate (Active Comparator): The intervention for this group is that the patient will undergo endoscopic ProTouch Laser Enucleation of Prostate (LEP).The laser is used to enucleate large pieces of prostatic tissue which is followed by further ablation of the tissue so that no fragments are left in the bladder
  Interventions: Procedure: ProTouch Laser Enucleation of Prostate (LEP)
- Transurethral Resection of Prostate (Active Comparator): The intervention for this group that the patient will undergo endoscopic Transurethral Resection of Prostate (TURP) using bipolar cautery. The prostate is essentially shaved down using sequential cuts and cautery.
  Interventions: Procedure: Transurethral Resection of Prostate (TURP)

INTERVENTIONS:
Procedure: ProTouch Laser Enucleation of Prostate (LEP) — Laser enucleation of the prostate is a standard form of treatment for BPH used widely. The ProTouch laser is established to be safe and is newer than the holmium laser.
  Arms: ProTouch Laser Enucleation of Prostate
Procedure: Transurethral Resection of Prostate (TURP) — TURP has been considered a gold standard for treatment of BPH in which rigid resectoscopes with bipolar cautery are used to endoscopically resect prostatic tissue.
  Arms: Transurethral Resection of Prostate

SUMMARY:
Benign prostatic hyperplasia (BPH) refers to the proliferation of smooth muscle and epithelial cells of the prostate gland. The enlarged gland has the potential to result in lower urinary tract symptoms (LUTS) secondary to either bladder outlet obstruction or increased muscle tone and resistance, or both.

For decades transurethral resection of the prostate (TURP) has been the gold standard for treatment of symptomatic BPH that is refractory to nonoperative management. This is a surgical intervention aimed to reduce the size of the prostate gland. However, over the past fifteen years, many alternative therapies have been introduced including laser enucleation of the prostate (LEP). LEP has numerous advantages including decreased blood loss and length of hospital stay as well as increased effectiveness and safety for large prostate gland sizes (>80g).

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of TURP to LEP using the ProTouch laser technology. While TURP has historically been the gold standard, LEP has become more widespread and is arguably a safer and more effective therapy for the patient. TURP is still widely performed because it is a traditional therapy with decades of data to support its efficacy, despite higher volume of blood loss and risk for TUR syndrome. In comparison, there is some data demonstrating that Holmium Laser Enucleation of the Prostate can have similar efficacy but may have longer operative times. The ProTouch laser is comparable to the Holmium laser but additionally provides improved hemostasis and tissue vaporization. There is little to no data comparing LEP with the ProTouch laser to TURP. This study will directly compare the efficacy of these two treatment methods by enrolling eligible subjects and comparing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age > 50-80 years
* Prostate gland size 50-100g
* Failure of nonoperative therapy
* IPSS 8+
* FR <15ml/s
* PVR <250
* If PVR is 250-400 then pre-operative urodynamics will be indicated
* Language: English, Spanish, Haitian Creole, French, Portuguese
* Willing to randomize

Exclusion Criteria:

* Neurogenic bladder
* PVR >400ml
* IPSS <8
* FR >15ml/Indwelling catheter

  - History of prostate cancer
* History of urethral stricture or vesicourethral anastomotic stricture
* Unable to be placed in lithotomy position
* Unable to undergo general or spinal anesthesia
* Unable to consent
* Untreated or uncorrected coagulopathy

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Urinary Flow Rate | From time of randomization and ultimately at 24 months
  Velocity (in cc/sec) of the urine flow

SECONDARY OUTCOMES:
Quality of Life score | From time of randomization and ultimately at 24 months
  Survey to determine how satisfied the patient is with urination
Blood loss | During surgery (full length of operative time)
  Amount of blood loss during surgery.
Catheter time | From time of surgery to up to 3 weeks after surgery.
  the amount of time a catheter must stay in place postoperatively
Post void residual | From time of randomization and ultimately at 24 months
  Amount of urine remaining in the bladder after voiding
Sexual Health Inventory for Men (SHIM) | From time of randomization and ultimately at 24 months
  Survey to assess baseline sexual function and whether this is affected by intervention type

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Wason, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No